CLINICAL TRIAL: NCT04998318
Title: Compare the Performance of the Pocket Colposcope to VIA/VILI for Triage of HPV+ Women in Kenya
Brief Title: 1:1 Comparison of the Pocket Colposcope in Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Kenya Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00106169
Record Dates: First submitted 2021-08-02; First posted 2021-08-10 (Actual); Results first posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Cervical Cancer; HPV Infection; HIV Infections
Keywords: cervical cancer screening, Pap smear, Colposcopy; Pap smear; colposcopy
MeSH Terms: conditions — Uterine Cervical Neoplasms; Papillomavirus Infections; HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard of Care (Active Comparator): Visual Inspection with Acetic Acid (VIA): First, the cervix should be wiped with a cotton swab to remove any preexisting mucous and/or blood. A 3-5% acetic acid solution will be applied to the cervix using a spray bottle or fox swab. After approximately 1-minute, any changes to the cervix using the naked eye will be noted. Acetic acid may be reapplied if acetowhitening diminishes during visual inspection.
  Visual Inspection with Lugol's Iodine (VILI): After imaging with Acetic acid, Lugol's iodine will be applied using a fox swab noting any yellow or non-staining areas. Lesion location(s) will be noted on a clock-face diagram and used to direct biopsy if a lesion is present or random biopsies will be obtained from two quadrants in the absence of a visible lesion.
  Interventions: Procedure: Standard of Care Colposcopy
- Pocket Colposcope (Experimental): Pocket-Assisted Visual Inspection with Acetic Acid (PA-VIA): The cervix should be wiped with a cotton swab to remove any preexisting mucous and/or blood. A 3-5% acetic acid solution will be applied using a spray bottle or fox swab. After approximately 1-minute, using the Pocket Colposcope any changes to the cervix will be noted. Using the Calla Health image acquisition software, both white and green images of the cervix will be captured at low-resolution. High-resolution green light images will be obtained at the provider's discretion. Acetic acid may be reapplied between white and green imaging at the provider's discretion if acetowhitening diminishes.
  Pocket-Assisted Visual Inspection with Lugol's Iodine (PA-VILI): After imaging with AA, Lugol's iodine will be applied using a fox swab noting any yellow or non-staining areas. Images will be acquired. A biopsy will be obtained using the pocket. Random biopsies will be obtained from 2 quadrants in the absence of a visible lesion.
  Interventions: Device: Pocket Colposcope

INTERVENTIONS:
Device: Pocket Colposcope — Both arms will receive treatment in order to prevent cervical cancer. However, the intervention using the pocket colposcope device will be used on half the enrolled subjects.
  Arms: Pocket Colposcope
Procedure: Standard of Care Colposcopy — VIA and VILI as previously described,
  Arms: Standard of Care

SUMMARY:
The Pocket colposcope has 510k FDA clearance and has been successfully used in almost 1500 unique patients globally in Duke and non-Duke protocols to date. 400 women who are HPV-positive and planned to undergo treatment at 6 Ministry of Health-supported outpatient clinics in Kisumu County will be recruited to the study. After providing informed consent, participants will be randomized 1:1 to either standard-of-care visual inspection or colposcopy with the Pocket Colposcope

DETAILED DESCRIPTION:
Women randomized to the standard-of-care arm will undergo VIA followed by Visual Inspection with Lugol's Iodine (VILI). Women randomized to the Pocket Colposcope arm will undergo Pocket-Assisted VIA (PA-VIA), green light imaging, and VILI using the Pocket Colposcope. Women in both arms will have biopsies taken of any suspicious lesions, or two biopsies taken in random locations if no lesions are visible. The locations of the biopsies will be based on provider impression. After their study-exams and biopsies are taken, women who are eligible for ablative treatment will be immediately treated in the clinic. Those with larger lesions or lesions concerning for invasive cancer will be referred to the local hospital for an excisional procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 25 years old and < 65 years old
2. Sex: Female
3. Positive HPV test within past 6 months
4. HIV+ women

Exclusion Criteria:

1. Pregnant women (cannot perform a cervical biopsy on a patient who is pregnant unless absolutely indicated)
2. Women with a negative HPV test
3. Patients incapable of giving informed consent
4. Women with a history of cervical cancer
5. Pelvic exam concerning for cervical cancer or cervical infection

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 434 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan Huchko, MD, Principal Investigator — Duke University
Locations (1):
- Kenya Medical Research Institute, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Pocket Colposcope; Mis-weighted Randomization to Pocket Colposcope: Pocket-Assisted Visual Inspection with Acetic Acid (PA-VIA): The cervix should be wiped with a cotton swab to remove any preexisting mucous and/or blood. A 3-5% acetic acid solution will be applied using a spray bottle or fox swab. After approximately 1-minute, using the Pocket Colposcope any changes to the cervix will be noted. Using the Calla Health image acquisition software, both white and green images of the cervix will be captured at low-resolution. High-resolution green light images will be obtained at the provider's discretion. Acetic acid may be reapplied between white and green imaging at the provider's discretion if acetowhitening diminishes.
- Standard of Care (VIA); Mis-weighted Randomization to Standard of Care (VIA): Visual Inspection with Acetic Acid (VIA): First, the cervix should be wiped with a cotton swab to remove any preexisting mucous and/or blood. A 3-5% acetic acid solution will be applied to the cervix using a spray bottle or fox swab. After approximately 1-minute, any changes to the cervix using the naked eye will be noted. Acetic acid may be reapplied if acetowhitening diminishes during visual inspection.
Period: Overall Study
Arm/Group | Pocket Colposcope | Standard of Care (VIA) | Mis-weighted Randomization to Pocket Colposcope | Mis-weighted Randomization to Standard of Care (VIA)
Started | 196 | 208 | 11 | 19
Completed | 196 | 197 | 11 | 19
Not Completed | 0 | 11 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pocket Colposcope | Standard of Care (VIA) | Mis-weighted Randomization to Pocket Colposcope | Mis-weighted Randomization to Standard of Care (VIA) | Total
Number analyzed (Participants) | 196 | 208 | 11 | 19 | 434
Age, Customized [Count of Participants; unit: Participants]
  25-34 years old | 49 | 56 | 2 | 3 | 110
  35-44 years old | 87 | 81 | 2 | 6 | 176
  45-54 years old | 45 | 46 | 5 | 8 | 104
  55-65 years old | 15 | 25 | 2 | 2 | 44
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 196 | 208 | 11 | 19 | 434
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 196 | 208 | 0 | 0 | 404
  Unknown or Not Reported | 0 | 0 | 11 | 19 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 196 | 208 | 11 | 19 | 434
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  Kenya | 196 | 208 | 11 | 19 | 434

OUTCOME MEASURES:

1. Primary Outcome: Percent of Exams With Lesions Identified
Description: The primary endpoint was the diagnostic accuracy of VIA versus the Pocket Colposcope for detecting CIN2+ lesions.
Time Frame: Baseline
Population: Participants who completed the study
Measure: Number (95% Confidence Interval); unit: percent of exams
Units Other Than Participants: Exams
Arm/Group | Pocket Colposcope | Standard of Care (VIA) | Mis-weighted Randomization to Pocket Colposcope | Mis-weighted Randomization to Standard of Care (VIA)
Number analyzed (Participants) | 196 | 197 | 11 | 19
Number analyzed (Exams) | 196 | 197 | 11 | 19
percent of exams | 14.3 [9.7 to 20.0] | 17.3 [12.4 to 23.1] | 0 [0 to 0] | 21.1 [2.3 to 39.8]

2. Primary Outcome: Sensitivity
Description: Sensitivity of Pocket vs VIA
Time Frame: Baseline
Population: Participants with biopsy results
Measure: Number; unit: percent
Arm/Group | Pocket Colposcope | Standard of Care (VIA)
Number analyzed (Participants) | 196 | 197
percent | 26.3 | 25.0

3. Primary Outcome: Specificity
Description: Specificity of Pocket vs VIA
Time Frame: Baseline
Population: Participants with biopsy results
Measure: Number; unit: percent
Arm/Group | Pocket Colposcope | Standard of Care (VIA)
Number analyzed (Participants) | 196 | 197
percent | 88.9 | 84.0

4. Primary Outcome: Negative Predictive Value (NPV)
Description: Negative predictive value (NPV) of Pocket vs VIA
Time Frame: Baseline
Population: Participants with biopsy results
Measure: Number; unit: percentage
Arm/Group | Pocket Colposcope | Standard of Care (VIA)
Number analyzed (Participants) | 196 | 197
percentage | 82.9 | 87.1

5. Primary Outcome: Positive Predictive Value (PPV)
Description: Positive predictive value (PPV) of Pocket vs VIA
Time Frame: Baseline
Population: Participants with biopsy results
Measure: Number; unit: percentage
Arm/Group | Pocket Colposcope | Standard of Care (VIA)
Number analyzed (Participants) | 196 | 197
percentage | 37.5 | 20.6

6. Secondary Outcome: Percent of Participants Who Reported Having No Awareness About Cervical Cancer and Cervical Cancer Prevention, Assessed by Questionnaire
Description: Participants were asked how much they knew about cervical cancer and cervical cancer prevention prior to the exam and after the visit.
Time Frame: baseline
Population: Participants who completed the questionnaire. Questionnaire data were not collected for the two mis-weighted randomization arms due to a lengthy enrollment pause prior to those arms being enrolled, as well as the randomization error. No data were collected from participants in the mis-weighted randomization arms, and there is no data to report.
Measure: Number; unit: percent of participants
Arm/Group | Pocket Colposcope | Standard of Care (VIA)
Number analyzed (Participants) | 190 | 197
percent of participants
  Pre-exam | 21.6 | 21.8
  Post-exam | 0.5 | 0.5

7. Secondary Outcome: Percent of Providers Who Reported Experiencing no Challenges During the Exam
Description: Providers perspective was assessed using the question: 'Did you run into any of the following challenges during today's exam?'.
Time Frame: baseline
Population: Provider surveys for participants who completed the study. Provider survey data were not collected for the two mis-weighted randomization arms due to a lengthy enrollment pause prior to those arms being enrolled, as well as the randomization error. No data were collected from participants in the mis-weighted randomization arms, and there is no data to report.
Measure: Number; unit: percent
Arm/Group | Pocket Colposcope | Standard of Care (VIA)
Number analyzed (Participants) | 191 | 197
percent | 96.3 | 97.0

8. Secondary Outcome: Percent of Participants Who Reported Experiencing Pain During Their Exam
Description: Participant perspective of the exam was assessed by asking "Did you experience any pain throughout your exam?"
Time Frame: Baseline
Population: as for outcome 6
Measure: Number; unit: percent of participants
Arm/Group | Pocket Colposcope | Standard of Care (VIA)
Number analyzed (Participants) | 190 | 197
percent of participants
  None | 21.6 | 21.8
  A little | 73.2 | 74.1
  Somewhat | 5.3 | 3.0
  Very much | 0 | 1.0

9. Secondary Outcome: Percent of Participants Who Expressed Confidence in Their Provider's Assessment
Description: Participant perspective of the exam was assessed by asking "How confident are you in the provider's assessment from today's visit?"
Time Frame: Baseline
Population: as for outcome 6
Measure: Number; unit: percent of participants
Arm/Group | Pocket Colposcope | Standard of Care (VIA)
Number analyzed (Participants) | 190 | 197
percent of participants
  None | 0.0 | 0.0
  A little | 3.2 | 2.5
  Somewhat | 28.4 | 28.4
  Very much | 68.4 | 69.0

10. Secondary Outcome: Percent of Participants Who Would Recommend the Exam to a Friend
Description: Participant perspective of the exam was assessed by asking "How likely would you recommend this medical exam to a friend?"
Time Frame: Baseline
Population: as for outcome 6
Measure: Number; unit: percent of participants
Arm/Group | Pocket Colposcope | Standard of Care (VIA)
Number analyzed (Participants) | 190 | 197
percent of participants
  Not likely at all | 0.0 | 0.5
  Not likely | 1.1 | 0.0
  Likely | 22.6 | 18.8
  Very likely | 76.3 | 80.7

ADVERSE EVENTS:
Time Frame: During baseline visit
Arm/Group | Pocket Colposcope | Standard of Care (VIA) | Mis-weighted Randomization to Pocket Colposcope | Mis-weighted Randomization to Standard of Care (VIA)
All-Cause Mortality (participants affected / at risk) | 0/196 | 0/208 | 0/11 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/196 | 0/208 | 0/11 | 0/19
Other Adverse Events (participants affected / at risk) | 0/196 | 0/208 | 0/11 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-03): https://cdn.clinicaltrials.gov/large-docs/18/NCT04998318/Prot_SAP_001.pdf